CLINICAL TRIAL: NCT03598946
Title: Evaluation of the Impact of a Screening Strategy Based on a Home Urinary Test in Non-respondent Women on a First Invitation to Papillomavirus Screening, on the Participation Rate Compared to a Uterine Cervix Smear Screening, With Taking Into Account the Socio-economic Level, During the Organized Screening for Cervical Cancer in Brittany
Brief Title: Urinary Human Papilloma Virus Test in the General Population in Brittany
Acronym: PapU-Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Association for the Screening of Cancers in Finistère (Other); ADECI35 (Unknown); ADECARMOR (Unknown); ADECAM INDUSTRIE (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC18.0092_PapU-Access
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Neoplasms,Ovarian
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Antibody-Coated Bacteria Test, Urinary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human Papilloma Virus Test urinary (Experimental): Urinary Test by a kit which is send to the woman's house
  Interventions: Device: Urinary test

INTERVENTIONS:
Device: Urinary test — Women use a home urinary test themselves

SUMMARY:
This is a population-based, prospective, multicenter and open-label study. 12,500 female non-respondents to the uterine cervix smear from 30 to 65 years of age in the context of the organized cervical cancer screening of the uterus, in the 4 Breton departments, will be proposed after stratification by age and socio-economic level at the revival of the cervical cancer of the uterus screening by the structure of management of Rennes, an invitation to the Human Papilloma Virus urine test thanks to the sampling kit sent to the home. It is planned a revival by simple mail after 4 months in one woman out of two who did not respond to this invitation to assess the impact of a recovery. This group represents about 5% of the eligible population in Brittany. The specimen will be sent by post with the signed consent and a questionnaire to the Hospital of Brest in virology laboratory for the detection of Human Papilloma Virus DNA (QPCR) in the urine (HPU test) and typing (LipA). In the case of a positive Human Papilloma Virus test, the woman being tested has a strong incentive to do the cervical cancer of the uterus with her doctor or midwife. In the case of abnormal smear, follow-up continues according to national recommendations to a gynecologist. All the data is collected on a software from the LINKS company, with the networking of the 4 Breton centers, the virology laboratory, and the Anatomy-Cytology-Pathology laboratories in Brittany; this collection will allow after extraction, a statistical analysis of the data. The analysis of the participation rate in this new screening, for each level of the socio-economic level, will allow a comparison with the participation in smear's revival of organized screening, between women's groups according to the socio-economic level of their residential place.

The project will take place over 24 months in 3 phases:

1. D0-M6: Pre-inclusion phase with implementation of the protocol (regulatory procedures, production of newsletters, consent, questionnaire, preparation of urine collection kits, postal validation).
2. M6-M18: Inclusion phase with start of the study, sending invitations and inclusion, Human Papillomavirus Urinary testing and uterine cervix smear monitoring.
3. M18-M24: Post-inclusion phase with assessment of the inclusions on the 4 Breton departments, verification and analysis of the data according to the socio-economic level, recovery of the uterine cervix smear stimulus data, realization of the statistical analyzes and budget impact analysis, communications and publications.

ELIGIBILITY:
Inclusion Criteria:

* Women from 30 to 65 years old who did not do uterine cervix smear and who live in Brittany

Exclusion Criteria:

* Women under 30 years or over 65 years
* Women of 30-65 years who have responded to the uterine cervix smear invitation
* Women who have had an uterine cervix smear raise
* Women who have already had an uterine cervix smear within 3 years
* Women who had a total hysterectomy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12500 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-10-29 (Estimated); Study Completion 2023-10-29 (Estimated)

PRIMARY OUTCOMES:
Rate of participation in the urinary group | 18 months
  To evaluate the rate of participation in the urinary test group

SECONDARY OUTCOMES:
Participation rate by different parameters | 18 months
  To evaluate the participation rate
Evaluation of access of the medical network with different indicators | 18 months
  To evaluate the access to the medical network
Evaluation of the Papillomavirus levels of genotype 16 and genotype 18 in the population | 18 months
  To evaluate the Papillomavirus levels of genotype 16 and genotype 18

CONTACTS AND LOCATIONS:
Locations (1):
- Christopher PAYAN, Brest, France

IPD SHARING:
Plan to Share IPD: No